CLINICAL TRIAL: NCT02308644
Title: Phase 3 Intravitreous Bevacizumab and Standard Metabolic Control for Diabetic Macular Edema - A Contrast Sensitivity Pilot Study.
Brief Title: Intravitreous Bevacizumab and Standard Metabolic Control for Diabetic Macular Edema - A Contrast Sensitivity Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Augusto Alves Lopes da Motta, Intravitreous Bevacizumab and standard metabolic control for Diabetic Macular Edema - A Contrast Sensitivity Study., University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 80838792A
Record Dates: First submitted 2014-11-24; First posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Retinopathy; intravitreal bevacizumab; Contrast Sensitivity
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Bevacizumab; Emergency Use Authorization

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab (Experimental): Group 1 - 21 eyes treated with intravitreal bevacizumab injection (1.25mg) at the weeks 0, 6,12 and 18 plus standard metabolic control with glycated hemoglobin measured at baseline, week 12 and 18. All patients were followed by expert (endocrinologist)
  Interventions: Drug: intravitreal bevacizumab injection(1.25mg)
- Sham (Sham Comparator): Group 2 - 20 eyes treated with sham injection at weeks 0 and 6; and intravitreal bevacizumab injection(1.25mg) in the weeks 12 and 18 plus standard metabolic control with glycated hemoglobin measured at baseline, week 12 and 18. All patients were followed by expert (endocrinologist)
  Interventions: Drug: intravitreal bevacizumab injection(1.25mg)

INTERVENTIONS:
Drug: intravitreal bevacizumab injection(1.25mg) — intravitreal bevacizumab injection(1.25mg) / Sham injection
  Other Names: Avastin, Genentech Inc., South San Francisco, CA, EUA

SUMMARY:
To evaluate the effects on contrast sensitivity (CS) measurements of intravitreal bevacizumab injections associated with standard metabolic control in eyes with diabetic macular edema (DME) associated with standard metabolic control.

DETAILED DESCRIPTION:
Prospective, randomized, masked and interventional study. Patients with diabetes mellitus (DM) 2, glycated hemoglobin (HbA1c) less than 11% and previously treated macular edema three months before will be randomized in two groups. The baseline examination consisted of visual acuity (VA), CS using the Pelli-Robson Charts, optical coherence tomography (OCT) and Fluorescein Angiography for all eyes.

The same tests will be repeated above, in both groups, again, in the week 2,6 and 12, when the data is then collected for analysis and so ended the closed phase. On the same day will start the open phase, which will be applied intravitreal injection of bevacizumab in both groups and the same tests of closed phase will be held in the week 14,18 and 24 when the study will be completed then [Table 1] .

Patients will be monitored and controlled clinically including blood pressure measurements, laboratory blood tests such as blood glucose, glycated hemoglobin, urea, creatinine, total cholesterol and fractions.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old, of both genders;
* Patients with diabetes mellitus type I or type II;
* Macular edema presence of clinically significant diabetic in their mixed or diffuse;
* Visual acuity worse than 20/40 corrected (< 68 letters ETDRS)
* Glycated hemoglobin ≤ 11%;
* Systolic and diastolic blood pressure < 170 and < 100 mmHg, respectively;
* Women not pregnant;
* Free and informed consent term signed the screening visit;
* Ability to adhere to the visits.

Exclusion Criteria:

* Failure to comply with any of the inclusion criteria;
* Treatment for DME within the prior 3 months;
* Vitreoretinal traction within 1 disc diameter (DD) of the fovea, clinically confirmed or with OCT;
* Atrophy or fibrosis surrounding the fovea;
* Any level of cataract;
* Vitreous hemorrhage or any opacity means;
* Eye disease related to diabetic retinopathy that can derail the central vision (eg Age Macula Degeneration, chorioretinitis scar, ...)
* Best-corrected visual acuity to 20/40 (> 68 letters ETDRS)
* Inability to understand the treatment and the term of consent;
* Debilitating systemic disorders that preclude the patient's admission to the study, according to the clinical judgment of the investigator;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Contrast sensitivity | 6 months (24 weeks )
  Evaluate the Contrast Sensitivity measured by Pelli-Robson charts (Clement Clarke Inc., Columbus, OH) at baseline, weeks 2,6,12,14,18 and 24 to be compared with visual acuity gold standard - Early Treatment of Diabetic Retinopathy Study - ETDRS charts

SECONDARY OUTCOMES:
Metabolic control | 6 months (24 weeks)
  Evaluate the effects of the standard metabolic control with glycated hemoglobin (HbA1c) levels in eyes with diabetic macular edema, measured by method certified by National Glycohemoglobin Standardization Program (NGSP) / reference values = 4.1 a 6.5%).

CONTACTS AND LOCATIONS:
Overall Officials: AUGUSTO MOTTA, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Motta AAL, Bonanomi MTBC, Ferraz DA, Preti RC, Sophie R, Abalem MF, Queiroz MS, Pimentel SLG, Takahashi WY, Damico FM. Short-term effects of intravitreal bevacizumab in contrast sensitivity of patients with diabetic macular edema and optimizing glycemic control. Diabetes Res Clin Pract. 2019 Mar;149:170-178. doi: 10.1016/j.diabres.2019.02.002. Epub 2019 Feb 11. PMID 30763599